CLINICAL TRIAL: NCT06235866
Title: Risk Identification of Long-term Complications in the Recover Patients With Severe COVID-19
Brief Title: Risk Identification of Long-term Complications
Status: Enrolling by invitation | Type: Observational
Sponsor: Wuhan Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20230922
Record Dates: First submitted 2023-10-08; First posted 2024-02-01 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Severe COVID-19
Keywords: COVID-19 Pneumonia; Long-term complications; Lung function
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Follow-up cohort of patients with severe COVID-19: The scores of various scales, pulmonary function and imaging changes of patients with severe COVID-19 were collected at 3 months, 6 months and 12 months after rehabilitation and discharge.
  Interventions: Other: Pulmonary rehabilitation

INTERVENTIONS:
Other: Pulmonary rehabilitation — According to the pulmonary rehabilitation guidelines, patients with severe COVID-19 were given regular rehabilitation treatment, including breathing exercises and physical rehabilitation exercises.

SUMMARY:
The investigators retrospectively analyze the clinical characteristics of severe COVID-19 in our hospital, and then establish a prediction model for long-term complications in patients with severe COVID-19, and strengthen follow-up to improve the prognosis of patients.

DETAILED DESCRIPTION:
At present, there is a lack of prediction models for the long-term complications of severe COVID-19. Therefore, the investigators used the hospital big data platform to retrospectively analyze the clinical characteristics of severe COVID-19 in our hospital, and conducted cohort follow-up of the changes in lung function including FEV1, FVC，FEV1% and DLCO, etc and and high-resolution CT of patients after discharge. COX model and other statistical methods were used to establish a prediction model for long-term complications of severe COVID-19, and early identification and intervention, strengthen follow-up, and improve the prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

The patient met the diagnostic criteria for severe COVID-19

Exclusion Criteria:

* Pregnant women Patients who died of COVID-19 Patients younger than 18 years of age without pulmonary CT

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with severe COVID-19 in our hospital from December 8, 2022 to January 31, 2023 were enrolled
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Lung function | 1 year
  Pulmonary function indicators improved gradually
Imaging of the lung | 1 year
  The residual lesions in the lung were gradually absorbed

CONTACTS AND LOCATIONS:
Locations (1):
- Follow-up of patients with severe COVID-19, Wuhan, China

IPD SHARING:
Plan to Share IPD: No
The project confidentiality agreement was observed, but the IPD could be made public after the study was completed.